CLINICAL TRIAL: NCT03867149
Title: Involvement of the Mediodorsal Nucleus of the Thalamus in Higher Order Cognitive Processes : a Study in Patients With a Thalamic Infarct
Brief Title: Involvement of the Mediodorsal Nucleus of the Thalamus in Higher Order Cognitive Processes
Acronym: THALEM2-0
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/18/0337; IDRCB (Other: 2018-A02779-46)
Record Dates: First submitted 2018-11-15; First posted 2019-03-07 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Thalamic Infarction
Keywords: Mediodorsal nucleus; higher order cognition
MeSH Terms: interventions — Neuroimaging; Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient with first thalamic infarct (Other): Patient with first thalamic infarct, they will undergo detailed neuropsychological assessment of memory, language, executive functions and mood along detailed neuroimaging including high-resolution imaging of the thalamus, DTI and resting state fMRI.
  Interventions: Other: neuroimaging; Other: Neuropsychological assessment
- healthy subject matched with control (Other): Healthy subject matched with control, they will undergo detailed neuropsychological assessment of memory, language, executive functions and mood along detailed neuroimaging including high-resolution imaging of the thalamus, DTI and resting state fMRI.
  Interventions: Other: neuroimaging; Other: Neuropsychological assessment

INTERVENTIONS:
Other: neuroimaging — neuroimaging including high-resolution imaging of the thalamus, DTI and resting state fMRI
Other: Neuropsychological assessment — neuropsychological assessment of memory, language, executive functions and mood

SUMMARY:
The aim is to expand evidence about the importance of the mediodorsal nucleus of the thalamus as a key node in human higher-order cognitive functions such as learning, decision-making, and adaptive behavior. Thus, the project proposes to assess global cognition along with higher-order cognition integrity via sensitive behavior tasks in patients with well localized lesions (mediodorsal thalamic infarcts) compared with healthy participants.

DETAILED DESCRIPTION:
The recruitment of patients with isolated thalamic lesion after stroke is known to be a challenge that the investigators overcame through the expertise of neurologists within their stroke unit.

First, they will describe the cognitive profile consecutive to a lesion of the thalamus, assessed with standardized neuropsychological tests.

Second, and more specifically, they will study performances at experimental tasks focusing on higher-order cognition (decision-making, updating, interference managing, multitasking).

They will use the automatic localization method already performed : the lesions will be manually segmented from T1 morphologic sequences, and then normalized in a template. Finally a numerical atlas of thalamus will be applied on the lesions, determining the injured substructure and the lesion volume.

Besides, this method will be compared with new high resolution thalamus-centered anatomical sequences allowing direct and individual identification of the involved thalamic nucleus.

ELIGIBILITY:
Inclusion criteria for patients:

* French as their mother tongue
* Absence of cognitive deterioration before the stroke.
* Visual, auditory (equipment authorized) and oral or written skills sufficient for the proper assessment using neuropsychological tests.
* First infarct affecting the thalamus.
* At least seven years' schooling from primary school
* Signed informed consent
* Chronic lesion (> 3 months)

Inclusion criteria for controls:

* French as their mother tongue
* Absence of cognitive complain
* Visual, auditory (equipment authorized) and oral or written skills sufficient for the proper assessment using neuropsychological tests.
* At least seven years of school from primary school
* Signed informed consent

Exclusion criteria for patients:

* Neurological deficit or significant residual disability at inclusion.
* Aphasia, agnosia, apraxia or severe neglect, as demonstrated by clinical examination and neuropsychological tests.
* Subjects with a contraindication to MRI.
* General, neurological or psychiatric progressive disease.

Exclusion criteria for controls:

* Subjects with a contraindication to MRI.
* General, neurological or psychiatric progressive disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-14 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Performance at the SET (Six Elements Test) | Day 1
  Performances of patients with a mediodorsal thalamic infarct in tasks assessing higher order cognition compared to healthy participants. Assessment of multitasking : 6 sub-tasks have to be achieved within 15 minutes.
  They include arithmetic tasks, image naming tasks, and dictation of a known route.
  Quantitative scores are derived from quantitative et qualitative data, then interpreted with international normative values.

SECONDARY OUTCOMES:
Performances at the PASAT (Pace Auditory Serial Addition Test) updating during working memory | Day 1
  Performances of patients with a mediodorsal thalamic infarct in sensitive executive tests compared to healthy participants.The PASAT assesses the updating during working memory.
Performances at the Brown-Petterson task | Day 1
  Performances of patients with a mediodorsal thalamic infarct in sensitive executive tests compared to healthy participants. The Brown-Petterson task focuses on the management of interference during working memory.

CONTACTS AND LOCATIONS:
Overall Officials: Jérémie PARIENTE, MD, PHD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Hopital Purpan - CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kopelman MD. What does a comparison of the alcoholic Korsakoff syndrome and thalamic infarction tell us about thalamic amnesia? Neurosci Biobehav Rev. 2015 Jul;54:46-56. doi: 10.1016/j.neubiorev.2014.08.014. Epub 2014 Sep 16. PMID 25218758
- [Background] Pergola G, Gunturkun O, Koch B, Schwarz M, Daum I, Suchan B. Recall deficits in stroke patients with thalamic lesions covary with damage to the parvocellular mediodorsal nucleus of the thalamus. Neuropsychologia. 2012 Aug;50(10):2477-91. doi: 10.1016/j.neuropsychologia.2012.06.019. Epub 2012 Jun 30. PMID 22750446
- [Background] Cipolotti L, Husain M, Crinion J, Bird CM, Khan SS, Losseff N, Howard RS, Leff AP. The role of the thalamus in amnesia: a tractography, high-resolution MRI and neuropsychological study. Neuropsychologia. 2008 Sep;46(11):2745-58. doi: 10.1016/j.neuropsychologia.2008.05.009. Epub 2008 May 21. PMID 18597798
- [Background] Danet L, Barbeau EJ, Eustache P, Planton M, Raposo N, Sibon I, Albucher JF, Bonneville F, Peran P, Pariente J. Thalamic amnesia after infarct: The role of the mammillothalamic tract and mediodorsal nucleus. Neurology. 2015 Dec 15;85(24):2107-15. doi: 10.1212/WNL.0000000000002226. Epub 2015 Nov 13. PMID 26567269